CLINICAL TRIAL: NCT06583837
Title: A Prospective, Multicenter, Phase II Study of Orelabrutinib Followed by Response-adapted Ultra-low Dose 4Gy Radiation as First-line Treatment of Local-stage Mucosa Associated Lymphoid Tissue Extranodal Marginal Zone Lymphoma
Brief Title: Orelabrutinib Followed by Response-adapted Ultra-low Dose 4Gy Radiation as First-line Treatment of MALT Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yizhen Liu, Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: iNHL-04
Record Dates: First submitted 2024-08-31; First posted 2024-09-04 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Lymphoma, B-Cell, Marginal Zone
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — orelabrutinib; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabrutinib followed by response-adapted ultra-low dose 4Gy radiation (Experimental): Orelabrutinib was administrated for 12 weeks, followed by response-adapted ultra-low dose 4Gy radiation for local stage MALT EMZL
  Interventions: Drug: Orelabrutinib; Radiation: response-adapted radiation

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib was administrated for 12 weeks
Radiation: response-adapted radiation — response-adapted ultra-low dose 4Gy radiation
  Other Names: radiation

SUMMARY:
Investigate the efficacy and safety of Orelabrutinib followed by response-adapted ultra-low dose 4Gy radiation in the treatment of local-stage MALT lymphoma

DETAILED DESCRIPTION:
This prospective, multicenter trial is trying to evaluate the efficacy and safety of Orelabrutinib followed by response-adapted ultra-low dose 4Gy radiation as first-line treatment of local-stage mucosa associated lymphoid tissue extranodal marginal zone lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Histologically confirmed mucosa-associated lymphoid tissue (MALT) lymphoma
* Lugano stage I-II
* ECOG 0-2
* Signed informed consent
* Having sufficient organ function: a) Hematopoietic function: Neutrophils ≥ 1.0 × 109/L, PLT ≥ 50 × 109/L, Hb ≥ 80g/L; b) Liver function: bilirubin ≤1.5 times the upper limit of normal (ULN), ALT and AST<3 x ULN, serum albumin ≥ 30 g/L; c) Renal function: serum Cr<1.5 × ULN, creatinine clearance rate ≥ 50mL/min (calculated according to the standard Cockcroft Gault formula, if renal dysfunction is caused by tumor compression, creatinine clearance rate ≥ 30mL/min); d) Coagulation function (unless the subject is receiving anticoagulant therapy and the coagulation parameters (PT/INR and APTT) are within the expected range of anticoagulant therapy at the time of screening): International standardized ratio (INR) ≤ 1.5 x ULN; Activated partial thromboplastin time (APTT) ≤ 1.5 x ULN.

Exclusion Criteria:

* Recent major surgery (within 4 weeks prior to enrollment), except for diagnostic surgery
* Have uncontrolled intercurrent diseases (cardiovascular and cerebrovascular diseases, coagulation disorders, severe infectious diseases) including but not limited to: severe acute or chronic infection requiring systemic treatment, symptomatic congestive heart failure (NYHA III-IV) or symptomatic or poorly controlled arrhythmias, arterial hypertension (systolic blood pressure ≥ 160mmHg or diastolic blood pressure ≥100mmHg) that is not controlled even with standard treatment, unstable angina, active peptic ulcer or bleeding disorder;
* Severe concomitant diseases that interfere with treatment
* Active interstitial pneumonia
* Active chronic hepatitis B infection (defined as HBV DNA positive; patients with latent or prior hepatitis B infection (defined as positive for hepatitis B surface antigen or hepatitis B core total antibody) can be included if HBV-DNA is undetectable at screening. The above-mentioned patients must voluntarily undergo regular DNA tests and receive appropriate antiviral therapy as prescribed)
* Positive hepatitis C test result (for patients who are positive for HCV antibodies, only polymerase chain reaction (PCR) shows a negative HCV RNA can participate)
* Patients with active HIV and syphilis infections;
* Pregnant or lactating women
* Patients with multiple factors affecting oral medication (such as dysphagia, nausea, vomiting, chronic diarrhea, and intestinal obstruction)
* The researcher determined that patients are not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
1-year event-free survival (EFS) | 1 year
  the period from the date of patients sign informed consent to the observed event for any reason

SECONDARY OUTCOMES:
6-months CR rate | up to 6 months
  the ratio of numbers of patients with complete response to all the participants receiving treatment
2-year event-free survival (EFS) | From date of patients sign informed consent until the date of first documented event, progression or date of death from any cause, whichever came first, assessed up to 2 years
  the period from the date of patients sign informed consent to the observed event for any reason
2-year progression-free survival (PFS) | From date of patients sign informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  the period from the date of patients sign informed consent to the observed progression of the disease or the occurrence of death for any reason
2-year overall survival rate | From date of patients sign informed consent until the date of death or the date of last follow-up time, whichever came first, assessed up to 2 years
  time between the date of patients sign informed consent and the date of death or the date of last follow-up time
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Throughout the treatment period, up to 1 year
  Record the name of adverse events and number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Quality of life questionnaire(EORTC QLQ-C30) | Up to 1 year
  evaluate patients' quality of life by questionnaire using EORTC QLQ-C30.There are a total of 30 entries. Among them, items 29 and 30 are divided into seven levels, ranging from 1 to 7 points based on their answer options; The other items are divided into four levels: none, a little, many to many, and are rated directly on a scale of 1 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China